CLINICAL TRIAL: NCT02485834
Title: Impact of Early FDG-PET Directed Intervention on Preoperative Therapy for Locally Advanced Gastric Cancer: A Random Assignment Phase II Study
Brief Title: FDG-PET Directed Treatment in Improving Response in Patients With Locally Advanced Stomach or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A021302; U10CA180821 (NIH); NCI-2014-02566 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Gastric Adenocarcinoma; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative; Fluorouracil; Capecitabine; Docetaxel; Irinotecan; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - surgery, chemotherapy and radiation therapy (Active Comparator): Patients undergo surgery within 42 days of completion of pre-registration chemotherapy. Beginning within 49 days of surgery, patients receive 5-FU IV continuously and capecitabine PO BID on days 1-7, and undergo 3D-CRT or IMRT QD on days 1-5. Treatment continues for 5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: surgery; Drug: 5-FU; Drug: capecitabine; Radiation: 3D-CRT; Radiation: IMRT
- Arm B - surgery, chemotherapy and FDG-PET (Experimental): Beginning within 28 days of day 1 of pre-registration chemotherapy, patients receive docetaxel IV and irinotecan IV on days 1 and 8. Treatment repeats every 3 weeks for 2 courses. Beginning within 42 days of completion of docetaxel and irinotecan, patients undergo surgery. Patients also undergo FDG-PET within 14 days of planned surgery. Beginning within 60 days after surgery, patients receive 3 additional courses of docetaxel and irinotecan hydrochloride courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: FDG-PET; Procedure: surgery; Drug: docetaxel; Drug: Irinotecan

INTERVENTIONS:
Procedure: FDG-PET
  Arms: Arm B - surgery, chemotherapy and FDG-PET
Procedure: surgery
Drug: 5-FU — 200 mg/m^2/day IV
  Arms: Arm A - surgery, chemotherapy and radiation therapy
Drug: capecitabine — oral 800 mg/m^2 BID
  Arms: Arm A - surgery, chemotherapy and radiation therapy
Drug: docetaxel — 30 mg/m^2 IV
  Arms: Arm B - surgery, chemotherapy and FDG-PET
Drug: Irinotecan — 50 mg/m^2 IV
  Arms: Arm B - surgery, chemotherapy and FDG-PET
Radiation: 3D-CRT
  Arms: Arm A - surgery, chemotherapy and radiation therapy
Radiation: IMRT
  Arms: Arm A - surgery, chemotherapy and radiation therapy

SUMMARY:
This randomized phase II trial studies how well fludeoxyglucose F-18 (FDG)/positron emission tomography (PET) directed treatment improves response in patients with stomach or gastroesophageal junction cancer that has not spread past the stomach and is not responding to the usual treatment. PET scans are a different way to take pictures of cancer and can be used to look at how much energy (such as glucose) is being used by the cancer. Using PET scans early to monitor the success of treatment may allow doctors to measure response and change treatment accordingly.

DETAILED DESCRIPTION:
Pre-registered patients receive standard pre-operative chemotherapy comprising epirubicin intravenously 50mg/m^2 (IV) on day 1; oxaliplatin 130 mg/m^2 IV or cisplatin 60 mg/m^2 IV on day 1; and capecitabine 625 mg/m^2 orally (PO) twice daily (BID) or fluorouracil 200 mg/m^2/day IV continuously on days 1-21; and undergo FDG-PET following course 1 (days 15-19). Patients defined as FDG-PET non-responders are registered and randomized to 1 of 2 treatment arms.

Primary objective

To assess and compare the overall survival (OS) of patients with locally advanced gastric cancer classified as FDG-PET non-responders after one cycle of pre-operative chemotherapy randomly assigned to receive either salvage chemotherapy before and after surgery or immediate surgery followed by fluorouracil sensitized radiotherapy.

Secondary objectives

1. To assess and compare progression-free survival (PFS) between the treatment arms (Arms A and B).
2. To assess and compare R0 resection rate between the treatment arms (Arms A and B).
3. To assess and compare pathologic complete response (pCR) rate between the treatment arms (Arms A and B).
4. To assess the adverse events (AE) profile and safety of each treatment arm (Arms A and B), including post-operative mortality rate, 30-day post-operative targeted adverse events (i.e., dehiscence, significant infection, and re-operation rate).
5. To examine the changes of FDG-PET SUV induced by pre-operative chemotherapy at different time points (from baseline to completion of one cycle of treatment before randomization, and 2 cycles of salvage treatment) in patients randomized to salvage treatment arm (Arm B).
6. To collect measurement of fatigue and overall perception of QOL at registration of the study (Alliance registration QOL assessment study).

ELIGIBILITY:
Pre-Registration Eligibility Criteria

1. Documentation of Disease

   1.1 Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (Siewert type II, III)

   1.2 Pre-treatment clinical stage of T3-4N any M0 or T any N positive M0 as determined by laparoscopy, CT scan (or PET/CT), or endoscopic ultrasound (histologic confirmation of lymph involvement is not required). Therefore, patients can have measurable or non-measurable disease.

   1.3 Patients with T1-2N0M0 tumors or patients with metastatic disease are NOT eligible.
2. Patients must be eligible for curative intent surgical resection.
3. FDG Avid malignancy - Patients must have an FDG avid tumor(s). FDG avid tumors are defined as a primary tumor with an increased uptake in the region of the tumor that has an SUV of > 5.0 or a tumor:liver SUV ratio of > 1.5.
4. No prior history of congestive heart failure - NYHA class I to IV or known DPD deficiency
5. No current grade 2, 3, or 4 of neuropathy.
6. No known hypersensitivity to epirubicin, oxaliplatin and cisplatin, capecitabine and 5-flurouracil, docetaxel or irinotecan.
7. Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects.

   7.1 Therefore, for women of childbearing potential only, a negative serum pregnancy test pregnancy test done ≤ 7 days prior to pre-registration is required.

   7.2 A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
8. Age ≥ 18 years
9. ECOG Performance Status 0 or 1
10. Required Initial Laboratory Values:

    * Absolute Neutrophil Count (ANC) ≥ 1,500/mm^3
    * Platelet Count ≥ 100,000/mm^3
    * Creatinine ≤ 1.5 x upper limit of normal (ULN)
    * Total Bilirubin ≤ 1.5 x ULN, except in patients with Gilbert's disease
    * AST and ALT ≤ 2.5 x ULN
    * Alkaline Phosphatase ≤ 2.5 x ULN

Registration Eligibility Criteria to Treatment Arms A or B

1. Patient must continue to be eligible for curative intent surgical resection.
2. Disease Progression: FDG avid malignancy that is classified as an FDG PET non- responder. PET non-responders are defined as having < 35% reduction in the FDG uptake of the primary tumor when compared to baseline.
3. Concomitant Medications -

   3.1 Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this trial. Patients on strong CYP3A4 inhibitors must discontinue the drug 14 days prior to the start of study treatment.

   3.2 Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment.
4. Patient must have received only one cycle of the following regimens during the pre-registration time period and no other therapy for gastric or gastroesophageal junction cancer:

   * Epirubicin, Oxaliplatin, and Capecitabine
   * Epirubicin, Oxaliplatin, and Fluorouracil
   * Epirubicin, Cisplatin, and Capecitabine
   * Epirubicin, Cisplatin, and Fluorouracil
5. Toxicity recovery should include the following:

   * Grade ≤ 2 neuropathy
   * Grade ≤ 2 diarrhea
   * Grade ≤ 2 mucositis
6. Pre-registration chemotherapy given within 42 days of treatment (treatment meaning surgery if Arm A, chemotherapy if Arm B)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, Study Chair — Weill Medical College of Cornell University
Locations (71):
- United States (71):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Saint Helena Hospital, St. Helena, California
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Kootenai Cancer Center, Post Falls, Idaho
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Freeman Health System, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pre-randomization events included: 1) Baseline FDG-PET scan 2) Pre-registration 3) Second FDG-PET scan. Screen failures excluded from the study before randomization consisted of ineligible patients (n = 13), investigator decision (n = 1), and other screen failure reason (n=1).
Period: Overall Study
Arm/Group | Arm A - Surgery, Chemotherapy and Radiation Therapy | Arm B - Surgery, Chemotherapy and FDG-PET
Started (Randomized) | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to small numbers, overall baseline characteristics are summarized across all randomized patients to protect patient confidentiality.
Groups:
- Randomized Patients: Patients on Arms A and B as detailed in the Participant Flow are summarized.
Arm/Group | Randomized Patients
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 3
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 3
    1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of randomization to death due to any cause.
Time Frame: Up to 3 years
Population: Due to small numbers, overall results are summarized across all randomized patients to protect patient confidentiality.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Patients
Number analyzed (Participants) | 5
months | NA [11.07 to NA] — Not all patients have observed event of interest (i.e. death); thus the median and upper 95% confidence interval limit are not available.

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Up to 3 years
Population: Due to small numbers, overall results are summarized across all randomized patients to protect patient confidentiality.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Patients
Number analyzed (Participants) | 5
months | NA [0.62 to NA] — Not all patients have observed event of interest (i.e. death/progression); thus the median and upper 95% confidence interval limit are not available.

3. Secondary Outcome: Number of Patients Achieved R0 Resection During Surgery
Description: The number of patients achieved R0 resection during surgery
Time Frame: At time of surgery
Population: Due to small numbers, overall results are summarized across all randomized patients to protect patient confidentiality.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Patients
Number analyzed (Participants) | 5
Participants | 3

4. Secondary Outcome: Number of Patients Had Pathologic Complete Response
Description: The number of patients had pathologic complete response (pCR). (pCR is defined as no gross or microscopic tumor identified with the surgical specimen. All lymph nodes should be free of tumor to document a PCR. If no gross tumor is visible, section around the area of inflammation (nodularity) should be made every 2-3 cm and specimens examined.)
Time Frame: Up to 3 years
Population: Due to small numbers, overall results are summarized across all randomized patients to protect patient confidentiality.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Patients
Number analyzed (Participants) | 5
Participants | 4

5. Secondary Outcome: Number of Participants Who Reported Grade 3 or Higher Adverse Events
Description: The number of patients who reported grade 3 or higher Adverse Events according to Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 30 days after completion of protocol treatment
Population: Only patients who received treatment and were assessed for adverse events and completed the adverse events form were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Patients
Number analyzed (Participants) | 4
Participants | 3

6. Other Pre Specified Outcome: Change in FDG-PET SUV Measures
Time Frame: Up to 14 days prior to surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are assessed prior to pre-registration, prior to registration, on day 1 of weeks 1 and 4 of chemo-radiation therapy for Arm A patients, on day 1 of each cycle (pre ad post-surgery) for Arm B patients, and prior to surgery for Arm A and B patients; Up to 30 days after completion of protocol treatment
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients assessed for AEs and completed AE form. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Arm A - Surgery, Chemotherapy and Radiation Therapy | Arm B - Surgery, Chemotherapy and FDG-PET
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Surgery, Chemotherapy and Radiation Therapy (N=2) | Arm B - Surgery, Chemotherapy and FDG-PET (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Surgery, Chemotherapy and Radiation Therapy (N=2) | Arm B - Surgery, Chemotherapy and FDG-PET (N=2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT02485834/Prot_SAP_000.pdf